CLINICAL TRIAL: NCT04405492
Title: Evaluation of Rapid Diagnostic Solutions, Serological and Molecular Tests for COVID-19
Acronym: ERap-COV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP200556
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV 2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Population 1 : Patients (Experimental): Hospitalized patients, positive or suspected of SARS-CoV-2 infection
  Interventions: Device: Taking blood samples (capillary and venous), saliva sampling and nasopharyngeal sampling.
- Population 2 : Hospital caregivers exposed to SARS-CoV-2 (Experimental): Longitudinal study of a hospital caregiver cohort
  Interventions: Device: Taking blood samples (capillary and venous), saliva sampling and nasopharyngeal sampling.
- Population 3 : Lay users (Experimental): Suitability of rapid test in view of its intended purpose for self-testing
  Interventions: Device: Capillary and salivary sampling

INTERVENTIONS:
Device: Taking blood samples (capillary and venous), saliva sampling and nasopharyngeal sampling. — After inclusion, demographic and medical data will be collected. Evaluated point-of-care devices will be tested immediately. Blood samples (capillary and venous), salivary sample and nasopharyngeal swab will be taken. Clinical samples will be stored in a dedicated biobank. Other SARS-CoV-2 diagnostic tests will be evaluated in the laboratory on the different clinical samples retrieved from the biobank.
  For all antigenic, molecular and serological tests evaluated, the reference method will be real-time RT-PCR as well as the result of medical imaging carried out as part of patient care.
  Arms: Population 1 : Patients
Device: Taking blood samples (capillary and venous), saliva sampling and nasopharyngeal sampling. — After inclusion, demographic and medical data will be collected. Point-of-care devices will be tested immediately. Blood samples (capillary and venous), salivary sample and nasopharyngeal swab will be taken (D0). A follow-up at D15, M1, M3, M6, M9 will be done. At each visit, participants will be asked information about their health status and their contacts with COVID-19 patients. Blood samples (capillary and venous), salivary sample and nasopharyngeal swab will be taken. Point-of-care devices will be tested during the visit.
  Cinical samples will be stored in a dedicated biobank. Other SARS-CoV-2 diagnostic tests will be evaluated in the laboratory on the different samples retrieved from the biobank.
  For all antigenic, molecular and serological tests evaluated, the reference method will be real-time RT-PCR as well as the result of medical imaging carried out as part of patient care.
  Arms: Population 2 : Hospital caregivers exposed to SARS-CoV-2
Device: Capillary and salivary sampling — Two rapid tests (NG Biotech) allowing anti-SRAS-CoV-2 antibodies detection from a fingerpick blood sample and antigen detection from a salivary sample will be provided in 3 pharmacies of Ile de France. The inclusion of lay persons will be carried out in pharmacies by investigators of the recruiting centers (Bacteriology and Virology departments). After inclusion, one of the tests will be given to the participant for self-testing. After performing the test, the participant will complete a questionnaire to give a feedback on the test usability and the result obtained.
  Arms: Population 3 : Lay users

SUMMARY:
Prospective study for clinical performance evaluation of COVID-19 diagnostic tests: detection of anti-SARS-CoV-2 antibodies by RDTs or ELISA (manual or automated), rapid diagnostic tests based on antigen detection, molecular or proteomic testing of SARS-CoV-2 (sensitivity, specificity, predictive values)

DETAILED DESCRIPTION:
Since initially reported in Wuhan, China, in late December 2019, the outbreak of SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) has spread globally, stressing many health systems especially intensive care unit (ICU) capacities thus resulting in high mortality. On 16 March 2020, WHO Director-General called on all countries to ramp up their testing programs as the best way to slow the advance of the coronavirus pandemic. Although the current gold standard for COVID-19 diagnosis remains real time reverse transcription-polymerase chain reaction (rRT-PCR), this technique has many shortcomings such as low sensitivity on nasopharyngeal swabs (70%). Multiple diagnostic test manufacturers have developed and begun selling rapid and easy-to-use devices. Before these tests can be recommended, they must be validated in the appropriate populations and settings.

Funded by French Defense Innovation Agency (AID), ERap-CoV is a prospective clinical study which aims to assess clinical performances of serological and antigenic assays for the diagnosis of SARS-CoV-2 infection, in comparison with current diagnostic tests on the market (immunological, proteomic, molecular). The ERap-CoV research will extend the clinical validation of the first NG-Test IgM-IgG COVID-19 point-of-care immunodiagnostic test (NG Biotech), which has shown excellent biological performance, compatible with the recommendations of the Haute Autorité de Santé (HAS) for serological assays (sensitivity> 90% and specificity> 98%, 15 days after symptoms) (1). Finally, AID funding will be used to develop 100% French-made serological and antigenic RDTs in less than a year.

ELIGIBILITY:
Common criteria for the 3 populations :

* Persons over 18 years of age
* Beneficiary or person entitled to a social security scheme

Population 1 (Patients) :

* Patients presenting for hospital admission on suspicion of SARS-Cov-2 infection based on the WHO definition and local guidelines
* Patient or relative/trusted person who has been informed about the study and has given informed consent.

Population 2 (Caregivers) :

* Caregivers exposed to COVID-19 in the course of their duties in the clinical departments of the Bicêtre and Paul Brousse hospitals.
* Caregiver who gave informed consent.

Population 3 (Lay Users) :

* Clients presenting themselves in one of the volunteer dispensary pharmacies located in the Île-de-France region, who will be called "lay users".
* Presentation on a study site

Exclusion Criteria:

Common criteria for the 3 populations:

- Person subject to a justice protection measure

Population 1 (Patients):

* Refusal to participate by the patient / support person or close friend
* Patient not speaking French and not accompanied by a translator
* Patient under guardianship or curatorship
* Person under AME (State medical aid)

Population 2 (Caregivers):

- Refusal to participate

Population 3 (lay users):

* Refusal to participate
* Person not speaking French and not accompanied by a translator
* Person under AME (State medical aid)
* Person out of state to consent, under guardianship or curatorship
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1210 (Estimated)
Dates: Start 2020-05-25 (Estimated); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of several diagnostic tests : tests based either on detection of the virus SARS-CoV-2 or detection of human antibodies generated in response to infection | Total duration of the study is 10 months
  * Tests based on detection of the virus SARS-CoV-2 (antigenic rapid tests, molecular tests, proteomic tests): sensibility and specificity compared to RT-PCR (Ct) in salivary samples and nasopharyngeal swabs from patients and cargivers included in the study
  * Tests based on detection of human antibodies generated in response to infection (rapid immunodiagnostic tests, ELISA): sensibility and specificity compared to RT-PCR (Ct) and ELISA (antibody titer) in blood or serum from patients and cargivers included in the study

SECONDARY OUTCOMES:
Sensitivity and specificity of immunological, antigenic, molecular and proteomic tests according to symptom duration, stage of the disease: asymptomatic, ambulatory, hospitalized, ventilated | Total duration of the study is 10 months
  Hospitalized patients, positive or suspected of SARS-CoV-2 infection are included in the study. Medical data related to COVID-19 infection will be recorded.
  Caregivers will be asked information about their health status related to a possible COVID-19 infection: symptoms if any, symptoms duration, severity.
Description of the incidence of infection among hospital caregivers, time to seroconversion according to clinical form, medium-term antibody persistence | Caregivers will be included in the study for 9 months. After inclusion (Day 0), follow-up visits at Day 15, 1 Month, 3 Months, 6 Months, 9 Months will be done.
  At each visit, participants will be asked information about their health status and their contacts with COVID-19 patients. Blood samples (capillary and venous), salivary sample and nasopharyngeal swab will be taken. Point-of-care devices will be tested during the visit.
Sensitivity and specificity of immunodiagnostic tests according to the sample used (serum and capillary blood) and according to the duration of the symptoms | Total duration of the study is 10 months
  Blood samples (capillary and venous) will be taken for serology testing from hospitalized patients, positive or suspected of SARS-CoV-2 infection and from hospital caregivers exposed to SARS-CoV-2. Participants will be asked information about their health status and medical data related to COVID-19 infection will be recorded.
Sensitivity and specificity of antigenic rapid tests, molecular tests, proteomic tests according to the sample used (salivary samples or nasopharyngeal swabs) and according to the duration of the symptoms | Total duration of the study is 10 months
  Blood samples (capillary and venous) will be taken for serology testing from hospitalized patients, positive or suspected of SARS-CoV-2 infection and from hospital caregivers exposed to SARS-CoV-2. Participants will be asked information about their health status and medical data related to COVID-19 infection will be recorded.
Suitability of rapid tests in view of its intended purpose for self-testing | 4 months
  Two rapid tests (NG Biotech) allowing anti-SRAS-CoV-2 antibodies detection from a fingerpick blood sample and antigen detection from a salivary sample will be provided in 3 pharmacies of Ile de France. The inclusion of lay persons will be carried out in pharmacies by investigators of the recruiting centers (Bacteriology and Virology departments). After inclusion, one of the tests will be given to the participant for self-testing. After performing the test, the participant will complete a questionnaire to give a feedback on the test usability and the result obtained.